CLINICAL TRIAL: NCT00829517
Title: Computer-Assisted Provision of Reproductive Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Eleanor Bimla Schwarz, Associate Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SFP2-8
Record Dates: First submitted 2009-01-23; First posted 2009-01-27 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Contraception; Sexually Transmitted Diseases
Keywords: Contraception; sexually transmitted diseases
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STI kiosk (Active Comparator): computer-assisted provision of screening for chlamydia
  Interventions: Other: STI module
- contraceptive kiosk (Experimental): computer-assisted provision of hormonal contraception
  Interventions: Other: computer-assisted provision of hormonal contraception

INTERVENTIONS:
Other: computer-assisted provision of hormonal contraception — a computer program available at a kiosk will offer women information about and a prescription for hormonal contraception that they can ask their clinician to sign.
  Other Names: Family planning kiosk
  Arms: contraceptive kiosk
Other: STI module — computer module available at a kiosk that will encourage women to be screened for chlamydia
  Other Names: Chlamydia kiosk
  Arms: STI kiosk

SUMMARY:
This project seeks to demonstrate that computer kiosks in a clinic waiting room can improve access to hormonal contraception and screening for sexually transmitted infections. The study will be a randomized controlled trial which will evaluate the use of a computer kiosk module to compare the proportion of women of reproductive age who receive a prescription for hormonal contraception when computer-assisted provision of hormonal contraception is offered (intervention) to encounters when the study clinic provides standard contraceptive care (control). Subjects will be contacted approximately 3 months (range 2-4 months) after the clinic visit to complete a follow-up phone interview. The study population will include English and Spanish-speaking women ages 18-45 who seek care at this clinic. Our hypothesis is that computer-assisted provision of hormonal contraception (intervention)will increase the proportion of women of reproductive age who receive a prescription for hormonal contraception versus standard contraceptive care(control).

DETAILED DESCRIPTION:
Data collection has been completed

ELIGIBILITY:
Inclusion Criteria:

* women who speak English or Spanish who visit a study clinic

Exclusion Criteria:

* women who do not speak English or Spanish

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 814 (Actual)
Dates: Start 2011-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
self-reported use of hormonal or more effective contraception | 3 months
receipt of screening for sexually transmitted infection | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor B Schwarz, MD, MS, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - UPMC, Pittsburgh, Pennsylvania